CLINICAL TRIAL: NCT02645526
Title: Is a Woolen Cap Effective in Maintaining Normothermia in Preterm Infants During Kangaroo Mother Care?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Padova (Other)
Collaborators: Doctors with Africa - Collegio Universitario Aspiranti Medici Missionari (CUAMM) (Unknown)
Responsible Party: Principal Investigator, Daniele Trevisanuto, MD, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUAMMcap
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Neonatal Temperature; Kangaroo Mother Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KMC with woolen cap (Experimental): In this group, the head of the patients will be covered with a woolen cap during KMC.
  Interventions: Other: Woolen cap
- KMC without woolen cap (No Intervention): In this group, the head of the patients will be uncovered during KMC.

INTERVENTIONS:
Other: Woolen cap
  Arms: KMC with woolen cap

SUMMARY:
The aim of the present study is to assess the effectiveness and the safety of a woolen cap in maintaining normothermia in low birth weight infants (LBWI) during Kangaroo Mother Care (KMC).

DETAILED DESCRIPTION:
Background: Neonatal hypothermia is an important challenge associated with morbidity and mortality. Preventing neonatal hypothermia is important in high resource countries, but is of fundamental importance in low resource settings where supportive care is limited.

Kangaroo mother care (KMC) is a low-cost intervention that, whenever possible, is strongly recommended for temperature maintenance. During KMC, the World Health Organization (WHO) guidelines recommend the use of a cap/hat, but its effect temperature control during KMC remains to be established.

In the hospitals participating to the projects of the non-governmental organization CUAMM, KMC represents a standard of care, but the head of the babies often remains uncovered due to local habits or to the unavailability of a cap.

Objective: The aim of the present study will be to assess the effectiveness and the safety of a woolen cap in maintaining normothermia in low birth weight infants (LBWI) during KMC.

Methods: This is a multicenter (three hospitals), multi country (three countries), prospective, unblinded, randomized clinical trial of KMC treatment with and without a woolen cap in LBWI. After obtaining parental consent, all infants with a birth weight <2500 g and candidate to KMC will be assigned to KMC with woolen cap or to KMC without cap group in a 1:1 ratio according to a computer-generated randomized sequence. The primary outcome measure will be the temperature in the normal range (36.5-37.5°C) in course of KMC during the first week of life. In all participants, axillary temperature will be measured with a digital thermometer 4 times per day. In addition, maternal and room temperature will be recorded. Secondary outcome measures will be: episodes of apnea; sepsis; mortality before hospital discharge; in-hospital growth; age at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight <2500 g (and)
* Candidate to KMC treatment (and)
* Parental consent; a written informed consent will be obtained by a member of the neonatal - Team involved in the study from a parent or guardian before KMC treatment

Exclusion Criteria:

* Major congenital malformations
* Twins
* Parental refusal to participate to the study

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Neonatal temperature in the normal range (36.5-37.5°C) in course of KMC treatment. | First week of life.

SECONDARY OUTCOMES:
Number of Participants With Sepsis defined as Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment. | Through study completion, an average of 2 weeks.
Number of participants died during hospital stay. | From date of randomization until the date of death from any cause, whichever came first, assessed up to 2 weeks.
Rate of growth (g/kg/die) during hospital stay. | From date of randomization until the date discharge,whichever came first, assessed up to 2 weeks.
Age at discharge. | From date of birth until the date discharge, whichever came first, assessed up to 2 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Daniele TREVISANUTO, Padua, IT-Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawn JE, Blencowe H, Oza S, You D, Lee AC, Waiswa P, Lalli M, Bhutta Z, Barros AJ, Christian P, Mathers C, Cousens SN; Lancet Every Newborn Study Group. Every Newborn: progress, priorities, and potential beyond survival. Lancet. 2014 Jul 12;384(9938):189-205. doi: 10.1016/S0140-6736(14)60496-7. Epub 2014 May 19. PMID 24853593
- [Background] Boundy EO, Dastjerdi R, Spiegelman D, Fawzi WW, Missmer SA, Lieberman E, Kajeepeta S, Wall S, Chan GJ. Kangaroo Mother Care and Neonatal Outcomes: A Meta-analysis. Pediatrics. 2016 Jan;137(1):e20152238. doi: 10.1542/peds.2015-2238. Epub 2015 Dec 23. PMID 26702029
- [Background] Lunze K, Hamer DH. Thermal protection of the newborn in resource-limited environments. J Perinatol. 2012 May;32(5):317-24. doi: 10.1038/jp.2012.11. Epub 2012 Mar 1. PMID 22382859
- [Background] Wyllie J, Bruinenberg J, Roehr CC, Rudiger M, Trevisanuto D, Urlesberger B. European Resuscitation Council Guidelines for Resuscitation 2015: Section 7. Resuscitation and support of transition of babies at birth. Resuscitation. 2015 Oct;95:249-63. doi: 10.1016/j.resuscitation.2015.07.029. Epub 2015 Oct 15. No abstract available. PMID 26477415
- [Derived] Cavallin F, Segafredo G, Pizzol D, Massavon W, Lusiani M, Wingi O, De Vivo M, Da Dalt L, Boscardin C, Manenti F, Putoto G, Trevisanuto D; CAP-KMC Group. Thermal Effect of a Woolen Cap in Low Birth Weight Infants During Kangaroo Care. Pediatrics. 2018 Jun;141(6):e20173073. doi: 10.1542/peds.2017-3073. Epub 2018 May 22. PMID 29789445
- [Derived] Trevisanuto D, Putoto G, Pizzol D, Serena T, Manenti F, Varano S, Urso E, Massavon W, Tsegaye A, Wingi O, Onapa E, Segafredo G, Cavallin F. Is a woolen cap effective in maintaining normothermia in low-birth-weight infants during kangaroo mother care? Study protocol for a randomized controlled trial. Trials. 2016 May 26;17(1):265. doi: 10.1186/s13063-016-1387-0. PMID 27229315